CLINICAL TRIAL: NCT05768646
Title: Counterfactual Thinking Assessment in Amyotrophic Lateral Sclerosis
Brief Title: Counterfactual Thinking in Amyotrophic Lateral Sclerosis
Acronym: CFTSLA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 23C122
Record Dates: First submitted 2023-02-22; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ALS patients
  Interventions: Behavioral: Neuropsychological instruments
- Healthy controls
  Interventions: Behavioral: Neuropsychological instruments

INTERVENTIONS:
Behavioral: Neuropsychological instruments — Neuropsychological instruments assessing cognitive (including counterfactual abilities), behavioural and psychopathological features

SUMMARY:
The properness of our past choices and action is usually judged according to what could have been if we had behaved differently. This ability to simulate alternatives to past factual events and actions is called counterfactual thinking (CFT) and is closely related to the decision-making process and future behaviors. In fact, the generation of CFT fulfills an important preparatory function, since it offers behavioral instructions that can guide the individual in facing similar decision-making problems in the future. Consequently, a damage or a reduction in the CFT are likely to impact on the individual's decision-making (DM) ability, especially regarding crucial decisions such as those in the medical field. In recent years, growing evidence has highlighted alterations in CFT in several neurological, neurodegenerative and psychiatric conditions, such as Huntington's disease, Parkinson's disease, prefrontal cortex damage, schizophrenia, obsessive-compulsive disorder and major depressive disorder, underlining how CFT deficits are specifically associated with frontal-executive dysfunction. These alterations, as mentioned, can lead to non-optimal DM processes and behaviors.

Amyotrophic Lateral Sclerosis (ALS) is a progressive neurodegenerative disease characterized by the loss of motor neurons in the spinal cord, brain stem and motor cortex. Literature data have highlighted the presence of cognitive and behavioral alterations as integral parts of the disease, as a part of a continuum, with a partial overlap, between ALS and frontotemporal dementia (FTD). The progressive and fatal course of the disease and the presence of cognitive/behavioral alterations, together with the impairment in communication skills, have significant implications on patient's competence in the advance care planning, especially regarding informed consent to advance treatment and end-of-life decision. In particular, patients' perspectives about therapeutic choices and end-of-life interventions are likely to be influenced by cognitive-behavioral aspects, where the integrity of frontal-executive functions plays a crucial role in patients' DM ability.

The investigators hypothesize that ALS patients will show a certain deficit in CFT, both in the ability to generate counterfactual thoughts related to a negative real-life and in the ability to use CFT to make causal inferences in fictional social scenarios. Moreover, a relationship between CFT and DM abilities is expected to be found. These expected impairments are likely to be associated with the cognitive and behavioral alterations that typically occur in ALS.

Primary aim The primary purpose of the study is to investigate the integrity of CFT ability in patients with ALS.

Specifically, this study aims to: (1) evaluate the functioning of the CFT in a group of patients affected by ALS; (2) investigate how the functioning of the CFT is associated with the ALS typical cognitive-behavioral alterations; (3) evaluate the possible association between CFT and DM abilities; (4) investigate how clinical, psychological, cognitive and behavioral variables affect CFT integrity.

Secondary aim CFT ability will be investigated along the course of the disease, with patients being recruited in a longitudinal study. When possible, according to clinical conditions, patients will be assessed at 0-6-12-24 months, in order to better characterize CFT and DM functioning over time, as well as patients' cognitive-behavioral profile. .

We expect to highlight a deficit or a reduction in patients' CFT ability and such alteration is likely to be associated with DM skills, as well as with the specific cognitive and behavioral profile of ALS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients: probable or definite ALS
* Healthy controls: not applicable

Exclusion Criteria:

* Patients: other brain disorders; severe general medical conditions and uncorrected visual/hearing deficits
* Healthy controls: brain disorders; severe general medical conditions and uncorrected visual/hearing deficits

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ALS patients coming to clinical attention and community resident healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 157 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Counterfactual Inference Test | At enrollment
  Performance-based tests assessing the ability to use CFT in order to make inferences
Spontaneous Counterfactual Generation Test | At enrollment
  Performance-based tests assessing CFT abilities, in particular the frequency of CFT generated in response to a personal, real-life event.

SECONDARY OUTCOMES:
Longitudinal assessment of CFT abilities | At enrollment
  Performance-based tests assessing the ability to use CFT in order to make inferences (i.e. Counterfactual Inference Test) and the frequency of CFT generated in response to a personal, real-life event (i.e., Spontaneous Counterfactual Generation Test) will be administered along the course of the disease, with patients being recruited in a longitudinal study. When possible, according to clinical conditions, patients will be assessed at 0-6-12-24 months, in order to better characterize CFT functioning over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy